CLINICAL TRIAL: NCT04712903
Title: A Phase IIIB, Single Arm Study, of Durvalumab in Combination With Platinum-Etoposide for Untreated Patients With Extensive-Stage Small Cell Lung Cancer Reflecting Real World Clinical Practice in Spain (CANTABRICO).
Brief Title: Durvalumab Plus Chemotherapy in Untreated Patients With Extensive-Stage Small Cell Lung Cancer
Acronym: CANTABRICO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D419QC00005; 2020-002328-35 (EudraCT Number)
Record Dates: First submitted 2020-12-03; First posted 2021-01-15 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Small Cell Lung Carcinoma Extensive Disease
Keywords: Extensive-Stage; ICI; SCLC; Durvalumab
MeSH Terms: interventions — durvalumab; Cisplatin; Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Durvalumab in Combination with Platinum-Etoposide (Experimental): Durvalumab 1500 mg via IV infusion will be concurrently administered with first-line chemotherapy (EP) on an every 3 week (q3w) schedule for 4 to 6 cycles, and will continue to be administered post-chemotherapy on an every 4 week (q4w) schedule until confirmed progressive disease (PD) or unacceptable toxicity.
  Interventions: Drug: Durvalumab; Drug: Cisplatin; Drug: Etoposide; Drug: Carboplatin

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg via IV infusion over 60 minutes on Day 1 of each cycle.
Drug: Cisplatin — Cisplatin as an IV infusion per local standards (usually over 60 to 120 minutes on Day 1) of each cycle.
Drug: Etoposide — Etoposide sequentially administered per local standards (usually over 30 to 60 minutes IV infusion) on Days 1, 2, and 3 of each cycle.
Drug: Carboplatin — Carboplatin as an IV infusion per local standards (usually over 30 to 60 minutes on Day 1) of each cycle.

SUMMARY:
This is a Phase IIIb, interventional, single arm, multicentre study to evaluate safety, effectivenees, use of resources and patient reporting outcomes in patients with ES-SCLC treated with durvalumab in combination with platinum-etoposide as first-line treatment in Spain.

DETAILED DESCRIPTION:
This trial will provide an opportunity to further evaluate the safety profile and efficacy of durvalumab + EP in patient population that is reflective of real-world clinical practice, Durvalumab will be concurrently administered with first-line chemotherapy (EP) on an every 3 week (q3w) schedule for 4 to 6 cycles, and will continue to be administered as monotherapy post-chemotherapy on an every 4 week (q4w) schedule until confirmed progressive disease (PD) or unacceptable toxicity.

Prophylactic cranial irradiation (PCI) is allowed in patients showing complete or partial responses after the durvalumab + EP combination cycles, at the discretion of the investigator according to their local clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented Small cell Lung Cancer with extensive disease.
* Patients who had received chemoradiotherapy for LS-SCLC and have experienced a treatment-free interval of at least 6 months since last chemotherapy, radiotherapy, or chemoradiotherapy cycle, can be included under investigator criteria.
* Brain metastases; must be asymptomatic or have been treated at least 2 weeks prior to study treatment and are currently receiving 10 mg/day or less of prednisone or equivalent.
* Patients must be considered suitable to receive a platinum-based chemotherapy regimen as 1st line treatment for ES-SCLC.
* ECOG Performance Status of 0-2 at enrolment.
* No prior exposure to immune-mediated therapy for cancer.
* Adequate hematologic and organ function.
* Life expectancy of at least 12 weeks.
* Body weight >30 kg.

Exclusion Criteria:

* Any history of radiotherapy to the chest prior to systemic therapy or planned consolidation chest radiation therapy (except paliative care outside of the chest).
* Paraneoplastic syndrome of autoimmune nature, requiring systemic treatment or clinical symptomatology suggesting worsening of PNS
* Active infection including tuberculosis, HIV, hepatitis B anc C
* Active or prior documented autoimmune or inflammatory disorders
* Uncontrolled intercurrent illness, including but not limited to interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Isla, M.D., Principal Investigator — Hospital Clínico Lozano Blesa, Zaragoza
Locations (28):
- Spain (28):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Badajoz
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Castellon
  - Research Site, Córdoba
  - Research Site, Galdakao
  - Research Site, Granada
  - Research Site, Jaén
  - Research Site, León
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Mataró
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Ourense
  - Research Site, Oviedo
  - Research Site, Palma
  - Research Site, Reus,Tarragona
  - Research Site, San Cristóbal de La Laguna
  - Research Site, San Sebastián
  - Research Site, Santander
  - Research Site, Santiago de Compostela
  - Research Site, Toledo
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Isla D, Zugazagoitia J, Arriola E, Garcia-Campelo R, Marti Blanco C, Diz-Tain MP, Lopez-Brea M, Moreno-Vega AL, Leon-Mateos L, Oramas J, Gutierrez-Calderon V, Majem M, Sanchez-Hernandez A, Aguado C, Alvarez-Cabellos R, Massuti B, Moreno A, Firvida-Perez JL, Valdivia J, Gonzalez-Cordero M, Zafra-Poves M, Domine M, Garcia-Navalon FJ, Villanueva N, Provencio M, Juan-Vidal O, Rivas-Corredor C, Olmedo Garcia ME, Palmero R, Lopez-Castro R, Carcereny E, Lechuga JL, Dominguez M, Callejo A, Paz-Ares L. Durvalumab plus platinum-etoposide in the first-line treatment of extensive-stage small cell lung cancer (CANTABRICO): A single-arm clinical trial. Lung Cancer. 2025 Nov;209:108763. doi: 10.1016/j.lungcan.2025.108763. Epub 2025 Sep 24. PMID 41033130
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00005&attachmentIdentifier=40fa9dfc-24d1-4222-8331-d930c6bb3390&fileName=D419QC00005_CSR_synopsis.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00005&attachmentIdentifier=901bd86a-a64f-4156-a1e8-0ed31672640b&fileName=D419QC00005_SAP.pdf&versionIdentifier=
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00005&attachmentIdentifier=2bd9ee06-7e52-491e-a204-58779ccf7f98&fileName=D419QC00005_Protocol.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 101 patients were included in the study have been analysed. All patients included in the analysis started treatment with chemotherapy and durvalumab and 81 of them started maintenance treatment with durvalumab.
Groups:
- Experimental Arm: Received study intervention
Period: Overall Study
Arm/Group | Experimental Arm
Started (101) | 101
Completed (101) | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: 101
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 80
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: Kg] | 75.6 (16.8)
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 46
  Former smoker | 53
  Not available | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs) Grade ≥ 3
Description: Patients with AEs grade ≥ 3 acording to NCI CTCAE v5.0
Time Frame: During study treatment, until disease progression (median 6 months)
Population: All patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Participants
  Yes | 77
  No | 24

2. Primary Outcome: Number of Patients With Immune-mediated Adverse Events (imAE)
Description: Patients with immune-mediated adverse events (imAE) per patient
Time Frame: During study treatment, until disease progression (median 6 months)
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental Arm: Received study treatment
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Participants
  Yes | 38
  No | 63

3. Secondary Outcome: Progression Free Survival (PFS).
Description: PFS: Defined as the time from the first date of treatment until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from investigational product or receives another anticancer therapy prior to progression. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable assessment.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Months | 6.1 [5.2 to 6.9]

4. Secondary Outcome: Objetive Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors (RECIST v1.0) Criteria for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: At least every 12 weeks, up to 18 monts
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Percentage of patients | 54.5 [44.7 to 64.2]

5. Secondary Outcome: Duration of Response (DoR)
Description: DoR: Defined as the time from the date of first documented response per RECIST1.1 until the first date of documented progression per RECIST1.1 or death in the absence of disease progression.
Time Frame: From the date of first documented response until the first date of documented progression or death in the absence of disease progression, assessed up to 2 years.
Population: Patients who achieved complete response or partial response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 55
Months | 5.6 [4.7 to 6.5]

6. Secondary Outcome: Time to Treatment Discontinuation (TTD)
Description: TTD: Defined as the time from the first date of treatment until the end of treatment date.
Time Frame: From the first date of treatment until the end of treatment date, assessed up to 2 years.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Months | 6.2 [4.5 to 9.9]

7. Secondary Outcome: Overal Survival (OS)
Description: OS: Defined as the time from the first date of treatment until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Time Frame: From date of inclusion until the date of death, assessed up to 30 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Months | 9.6 [7.8 to 11.3]

8. Secondary Outcome: PFS Rate at 6 Months
Description: Percentage of participants remaining alive without disease progression at 6 months after initiation of study treatment.
Time Frame: Every 12 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Percentage of patients | 53.0 [43.2 to 62.8]

9. Secondary Outcome: PFS Rate at 12 Months
Description: Percentage of participants remaining alive without disease progression at 12 months after initiation of study treatment.
Time Frame: Every 12 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Percentage of patients | 21.0 [13.0 to 29.0]

10. Secondary Outcome: DoR Rate at 12 Months
Description: Percentage of responders remaining alive without disease progression at 12 months after first response.
Time Frame: Every 12 weeks
Population: Patients who achieved complete response or partial response.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Experimental Arm
Number analyzed (Participants) | 55
Percentage of patients | 35.7 [23.0 to 48.4]

11. Secondary Outcome: OS Rate at 6 Months
Description: Percentage of participants remaining alive at 6 months after initiation of study treatment.
Time Frame: Every 12 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Percentage of patients | 75.2 [66.8 to 83.6]

12. Secondary Outcome: OS Rate at 12 Months
Description: Percentage of participants remaining alive at 12 months after initiation of study treatment.
Time Frame: Every 12 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Percentage of patients | 40.7 [31.1 to 50.3]

13. Secondary Outcome: OS Rate at 18 Months
Description: Percentage of participants remaining alive at 18 months after initiation of study treatment.
Time Frame: Every 12 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Experimental Arm
Number analyzed (Participants) | 101
Percentage of patients | 31.6 [22.4 to 40.8]

14. Secondary Outcome: EORTC QLQ-C30: Global Health Status Domain, Change From Baseline to End of Treatment Visit
Description: EORTC QLQ-C30 was administered on day 1 and on the final visit (last treatment visit). EORTC QLQ-C30 is a 30-item questionnaire used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status scale, 5 functional scales (Physical Functioning, Role Functioning, Cognitive Functioning, Emotional Functioning, Social Functioning), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrohea, Financial difficulties).
  For each of these scales, scores range from 0 to 100. For the Global Health Status and the 5 functional scales a high score indicates better global health status/functioning and a positive change from baseline indicates improvement.
  Change from baseline is the difference in the score between the end of treatment visit and the first visit.
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Completed: Completed the items in the questionnaire.
Arm/Group | Completed
Number analyzed (Participants) | 67
Units on a scale | -6.3 (30.8)

15. Secondary Outcome: EORTC QLQ-C30: Physical Functioning Domain, Change From Baseline to End of Treatment Visit
Description: as for outcome 14
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | -15.0 (29.4)

16. Secondary Outcome: EORTC QLQ-C30: Role Functioning Domain, Change From Baseline to End of Treatment Visit
Description: as for outcome 14
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | -17.0 (36.0)

17. Secondary Outcome: EORTC QLQ-C30: Emotional Functioning Domain, Change From Baseline to End of Treatment Visit
Description: as for outcome 14
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | -2.3 (30.4)

18. Secondary Outcome: EORTC QLQ-C30: Cognitive Functioning Domain, Change From Baseline to End of Treatment Visit
Description: as for outcome 14
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | -15.0 (24.0)

19. Secondary Outcome: EORTC QLQ-C30: Social Functioning Domain, Change From Baseline to End of Treatment Visit
Description: as for outcome 14
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 67
Units on a scale | -12.0 (31.0)

20. Secondary Outcome: EORTC QLQ-C30: Fatigue, Change From Baseline to End of Treatment Visit
Description: EORTC QLQ-C30 was administered on day 1 and on the final visit (last treatment visit). EORTC QLQ-C30 is a 30-item questionnaire used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical Functioning, Role Functioning, Cognitive Functioning, Emotional Functioning, Social Functioning), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrohea, Financial difficulties).
  For the 9 symptom scales, a high score indicates a higher level of symptoms, and a negative change from Baseline indicates an improvement in symptoms.
  Change from baseline is the difference in the score between the end of treatment visit and the first visit.
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | 12.4 (29.4)

21. Secondary Outcome: . EORTC QLQ-C30: Pain, Change From Baseline to End of Treatment Visit
Description: as for outcome 20
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | 0.2 (29.2)

22. Secondary Outcome: EORTC QLQ-C30: Nausea and Vomiting, Change From Baseline to End of Treatment Visit
Description: as for outcome 20
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | 0.7 (20.1)

23. Secondary Outcome: EORTC QLQ-C30: Dyspnoea, Change From Baseline to End of Treatment Visit
Description: as for outcome 20
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | -2.4 (37.2)

24. Secondary Outcome: EORTC QLQ-C30: Insomnia, Change From Baseline to End of Treatment Visit
Description: as for outcome 20
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 68
Units on a scale | 1.0 (36.4)

25. Secondary Outcome: EORTC QLQ-C30: Appetite Loss, Change From Baseline to End of Treatment Visit
Description: as for outcome 20
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | -2.4 (36.3)

26. Secondary Outcome: EORCT QLQ-C30: Constipation, Change From Baseline to End of Treatment Visit
Description: as for outcome 20
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | 6.3 (33.5)

27. Secondary Outcome: EORTC QLQ-C30: Diarrhoea, Change From Baseline to End of Treatment Visit
Description: as for outcome 20
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 69
Units on a scale | 0.0 (18.1)

28. Secondary Outcome: EORTC QLQ-C30: Financial Difficulties, Change From Baseline to End of Treatment Visit
Description: as for outcome 20
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 65
Units on a scale | 10.3 (22.0)

29. Secondary Outcome: EORTC QLQ-LC13: Coughing, Change From Baseline to End of Treatment Visit
Description: EORTC QLQ-LC13 is a 13-items questionnaire used in clinical research to assess health-related quality of life in lung cancer patients. The QLQ-LC13 includes questions assessing lung cancer-associated symptoms (Coughing, haemoptysis, dyspnoea and site specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy and alopecia) and pain medication.
  Scores are calculated and transformed to range from 0 to 100. For the disease symptoms and side-effects of treatment scales a higher score represents a higher level of symptoms/problems and a negative change from baseline value indicates reduction (i.e. improvement) in symptoms.
  Change from baseline is the difference in the score between the end of treatment visit and the first visit.
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 73
Units on a scale | -7.8 (29.7)

30. Secondary Outcome: EORTC QLQ-LC13: Haemoptysis, Change From Baseline to End of Treatment Visit
Description: as for outcome 29
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 73
Units on a scale | -0.5 (15.2)

31. Secondary Outcome: EORTC QLQ-LC13: Dyspnoea, Change From Baseline to End of Treatment Visit
Description: as for outcome 29
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 68
Units on a scale | 3.1 (24.1)

32. Secondary Outcome: EORTC QLQ-LC13: Pain in Arm or Shoulder, Change From Baseline to End of Treatment Visit
Description: as for outcome 29
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 71
Units on a scale | 3.3 (33.4)

33. Secondary Outcome: EORTC QLQ-LC13: Pain in Other Parts, Change From Baseline to End of Treatment Visit
Description: as for outcome 29
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 68
Units on a scale | 7.4 (39.4)

34. Secondary Outcome: EORTC QLQ-LC13: Sore Mouth, Change From Baseline to End of Treatment Visit
Description: as for outcome 29
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 71
Units on a scale | 2.3 (13.0)

35. Secondary Outcome: EORTC QLQ-LC13: Peripheral Neuropathy, Change From Baseline to End of Treatment Visit
Description: as for outcome 29
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 71
Units on a scale | 13.6 (27.4)

36. Secondary Outcome: EORTC QLQ-LC13: Alopecia, Change From Baseline to End of Treatment Visit
Description: as for outcome 29
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 72
Units on a scale | 18.1 (37.5)

37. Secondary Outcome: EORTC QLQ-LC13: Dysphagia, Change From Baseline to End of Treatment Visit
Description: as for outcome 29
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 72
Units on a scale | 2.8 (23.6)

38. Secondary Outcome: EORTC QLQ-LC13: Chest Pain Item Change From Baseline to End of Treatment Visit
Description: as for outcome 29
Time Frame: Baseline (cycle 1 day 1) and end of treatment visit.
Population: Enrolled participants who completed baseline and end of treatment questionnaires.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Completed
Number analyzed (Participants) | 73
Units on a scale | -1.8 (29.3)

ADVERSE EVENTS:
Time Frame: During study treatment, until disease progression (median 6 months)
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 76/101
Serious Adverse Events (participants affected / at risk) | 57/101
Other Adverse Events (participants affected / at risk) | 100/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=101)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (10)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (3)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2 (2)
Diplopia (Eye disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2)
Herpes zoster reactivation (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Radial head dislocation (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebellar syndrome (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Immune-mediated neurological disorder (Nervous system disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1)
Neurological decompensation (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (3)
Spinal cord compression (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1)
Renal tubular disorder (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (2)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=101)
Anaemia (Blood and lymphatic system disorders) | 50 (125)
Asthenia (General disorders) | 64 (157)
Neutropenia (Blood and lymphatic system disorders) | 34 (56)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (40)
Constipation (Gastrointestinal disorders) | 27 (35)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (31)
Diarrhoea (Gastrointestinal disorders) | 21 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (28)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (27)
Nausea (Gastrointestinal disorders) | 18 (22)
Decreased appetite (Metabolism and nutrition disorders) | 18 (19)
Pyrexia (General disorders) | 15 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (19)
Hypothyroidism (Endocrine disorders) | 15 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (23)
Vomiting (Gastrointestinal disorders) | 12 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (13)
Platelet count decreased (Investigations) | 11 (15)
Mucosal inflammation (General disorders) | 10 (12)
Respiratory tract infection (Infections and infestations) | 10 (12)
Urinary tract infection (Infections and infestations) | 9 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (13)
Oedema peripheral (General disorders) | 8 (13)
Neutrophil count decreased (Investigations) | 8 (15)
Headache (Nervous system disorders) | 8 (8)
Insomnia (Psychiatric disorders) | 8 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 8 (11)
Hyperthyroidism (Endocrine disorders) | 7 (8)
Alanine aminotransferase increased (Investigations) | 7 (10)
Amylase increased (Investigations) | 7 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Acute kidney injury (Renal and urinary disorders) | 6 (6)
Fatigue (General disorders) | 6 (10)
Illness (General disorders) | 6 (8)
COVID-19 (Infections and infestations) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 6 (9)
Dizziness (Nervous system disorders) | 5 (6)
Gamma-glutamyltransferase increased (Investigations) | 5 (11)
Lymphocyte count decreased (Investigations) | 5 (13)
Dysgeusia (Nervous system disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT04712903/Prot_004.pdf
  • Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT04712903/SAP_005.pdf